CLINICAL TRIAL: NCT06079190
Title: A Phase 2, Parallel Group, Randomized, Double- Blind, Placebo-Controlled, 3-Arm, Multicenter Treatment Study to Evaluate the Efficacy and Safety of GSK4527226 [AL101] Intravenous Infusion Compared With Placebo in Patients With Early Alzheimer's Disease
Brief Title: Efficacy and Safety of GSK4527226 [AL101] in Participants With Early Alzheimer's Disease
Acronym: PROGRESS-AD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Alector Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 219867; 2023-505083-11-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- GSK4527226 Dose 1 (Experimental): Participants will receive GSK4527226 Dose 1
  Interventions: Drug: GSK4527226
- GSK4527226 Dose 2 (Experimental): Participants will receive GSK4527226 Dose 2
  Interventions: Drug: GSK4527226
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK4527226 — GSK4527226 will be administered.
  Arms: GSK4527226 Dose 1; GSK4527226 Dose 2
Other: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
The aim of this study is to assess the efficacy and safety of GSK4527226 in participants with early Alzheimer's Disease (AD) (including mild cognitive impairment [MCI] and mild dementia due to AD) of 2 dose levels of GSK4527226 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

Participant must be in the Alzheimer's continuum as defined by the 2018 National Institute on Aging and Alzheimer's Association (NIAAA) Research Framework corresponding to the clinical categories of MCI due to AD and mild AD dementia.

Participant must have evidence of amyloid positivity either by positive positron emission tomography (PET) result (Amyloid PET scans must be read by a central imaging lab) or cerebrospinal fluid (CSF) amyloid beta (Aβ) test result indicative of amyloid positivity

* Participants must also meet the following criteria for clinical severity:

  1. MMSE score of between 21 and 29 points
  2. CDR-global score (GS) of 0.5 to 1.0.
  3. CDR Memory Box score greater than or equal to (≥) 0.5.
  4. Participants with objective impairment in episodic memory as indicated by at least 1 standard deviation below age-adjusted mean in the Wechsler Memory Scale-IV Logical Memory II (WMS-IV LMII)
* If the participant is receiving symptomatic AD medications such as an Acetylcholinesterase inhibitor (AChEI) or memantine, the dosing regimen must have been stable for at least 12 weeks prior to screening and is not expected to change during study participation.
* If the participant is receiving other medications for AD related symptoms or associated conditions, the dosing regimen must have been stable for at least 4 weeks prior to screening and not expected to change during study participation. Symptoms must be considered adequately and stably controlled by the investigator, without marked changes in medication anticipated for the duration of the study.
* Body weight ≥ 45 kilogram (kg) to less than or equal to (≤)120 kg with body mass index (BMI) between 17 and 34.9 kilogram per meter square (kg/m^2), inclusive.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and if of child-bearing potential follows contraception requirements outlined in the protocol
* A male participant is eligible to participate if he follows contraception requirements outlined in the protocol
* Willing and able to give informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
* Availability of an adult person who has frequent and sufficient contact with the participant is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits, and signs the ICF of the study partner.

Exclusion Criteria:

Participant has evidence of any neurological condition other than AD that may contribute to cognitive impairment.

* History or presence of vascular disease that has the potential to affect cognitive function.
* History or presence of stroke within the past 1 year or recent transient ischemic attack within 180 days before screening.
* History of severe, clinically significant central nervous system (CNS) trauma.
* History or presence of intracranial tumor.
* Presence of ongoing infection(s) that may affect brain function, or history of infections that resulted in neurologic sequelae.
* History of primary psychiatric diagnosis that the investigator considers may interfere with study assessments.

Columbia Suicide Severity Rating Scale (C-SSRS) suicidal ideation Type 4 or 5, suicidal behaviour or has been assessed to be at risk of suicide, in the opinion of the investigator within 6 months before screening, at screening, or at the Baseline visit, or has been hospitalized or treated for suicidal behaviour in the past 2 years.

* Participant has history of alcohol and/or moderate to severe substance use disorder within the past 2 years
* Magnetic resonance imaging (MRI) evidence based on central read of:

  1. >3 lacunar infarcts.
  2. Stroke involving a major vascular territory, severe small vessel, or white matter disease.
  3. Any territorial /cortical/other infarct >1 cubic centimetre (cm^3).
  4. White matter hyperintense lesions on the FLAIR sequence that correspond to an overall Fazekas score of 3
  5. >4 microhaemorrhages.
  6. Any areas of superficial (leptomeningeal) hemosiderosis.
  7. A single macro-hemorrhage greater than 10 millimetres (mm) at greatest diameter.
  8. Vasogenic edema.
  9. Cerebral contusion, encephalomalacia, aneurysms, vascular malformations, or infective lesions.
  10. Space occupying lesions or brain tumors.
  11. Significant cerebral vascular pathology
  12. Hydrocephalus/Normal pressure hydrocephalus.
  13. Other MRI findings contraindicating participation in the study such as subarachnoid hemorrhage.
* History suggestive of exposure to, or past tuberculosis (TB) infection should undergo screening for TB disease.
* Chronic active immune disorder requiring systemic immunosuppressive therapy within 6 months prior to Screening.
* Screening serum vitamin B12 concentration < Lower limit of normal (LLN) or in the low normal range
* Folate <LLN or Thyroid-stimulating hormone (TSH) > Upper limit of normal (ULN)
* Hemoglobin A1c >8 percentage (%) or poorly controlled diabetes during the last 12 weeks
* History of cancer
* Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human, or humanized antibodies or fusion proteins
* Planned surgery during the study which requires general, spinal, or epidural anesthesia that would take place during the study.
* Known genetic predisposition for clotting disorder or hemorrhagic disease.
* Key exclusionary medications include:

  * Antipsychotics, opiates/opioids, cannabinoids, hypnotics, antidepressants, mood stabilizers, or stimulants that are used on a chronic basis, are exclusionary if not consistent with the following rule: treatment has to have been at a stable dose for at least 4 weeks before screening and should remain stable during the study
  * Any biologic drugs with systemic exposure, whether investigational or approved, used within 6 months before screening Any disease modification drug for AD, such as aducanumab and lecanemab, whether investigational or approved, used within 6 months before screening.
  * Anticoagulation medications within 90 days of screening and during the study
  * Systemic immunosuppressive therapy within 6 months before screening and during the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) Score for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Week 52, 64 and 76
  The CDR-SB score is a quantitative general index that provides more precision in participants with mild dementia. The CDR scale is a clinician-rated dementia staging system tracks the progression of. cognitive impairment in 6 categories (memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5- point scale in which None=0, Questionable=0.5, Mild=1, Moderate=2, and Severe=3. The CDR-SB is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment.

SECONDARY OUTCOMES:
Change from Baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) Score for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Weeks 52, 64 and 76
  The iADRS is a composite score that measures both cognition and function. The iADRS comprises scores from the AD Assessment Scale-Cognitive subscale (ADAS-Cog) and the Alzheimers Disease Cooperative Study-instrumental Activities of Daily Living (ADCS-iADL). The iADRS is calculated as a linear combination of the total scores of the ADAS-Cog14 (14-item version of the test that assesses immediate and delayed memory, confrontational naming, ability to follow commands, ideational and constructional praxis, orientation, language, and attention. Higher scores indicate greater impairment) and the ADCS-iADL (score range from 0-49 with higher scores reflecting better performance and lower scores indicating greater functional impairment).
Change from Baseline in ADAS-Cog14 Score for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Weeks 52, 64 and 76
  The AD Assessment Scale-Cognitive subscale (ADAS-Cog14) is a 14-item version of the test that assesses immediate and delayed memory, confrontational naming, ability to follow commands, ideational and constructional praxis, orientation, language, and attention. Score ranges from 0 to 90 and higher scores indicate greater impairment.
Change from Baseline in ADCS-ADL-MCI Score for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Weeks 52, 64 and 76
  The AD Cooperative Study - Activities of Daily Living Scale for use in Mild Cognitive Impairment (ADCS-ADL-MCI). The ADCS-ADL for MCI is a 23-item scale that measures the competence of participants in basic and instrumental activities of daily living. Total scores on the ADCS-ADL-MCI range from 0 to 53 where lower scores indicates greater functional impairment.
Change from Baseline in ADCS-iADL component of ADCS-ADL-MCI Score for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Weeks 52, 64 and 76
  The ADCS-iADL is a subscale which measures instrumental activities of daily living. The ADCS-iADL is derived from the ADCS-ADL-MCI. It has a total score ranging from 0 to 49 with lower scores indicating greater functional impairment.
Change from Baseline in Alzheimer's Disease Composite Score (ADCOMS) for Dose 1 vs Placebo Across Weeks 52, 64 and 76 | Baseline, Weeks 52, 64 and 76
  The ADCOMS is a composite score comprising scores from various items of the Mini-Mental Status Examination (MMSE), ADAS-Cog14, and CDR domains. The MMSE is a brief test used to screen for cognitive impairment. It is routinely used for estimating the severity of cognitive impairment and tracking cognitive changes in an individual over time. It assesses orientation (time and place), registration, attention and calculation, recent memory, language (naming, comprehension, and repetition), and constructional praxis (copying a figure). For ADCOMS a higher score is indicative of greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (86):
- United States (19):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Lake Mary, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, The Villages, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Chesterfield, Missouri
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Matthews, North Carolina
  - GSK Investigational Site, North Canton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Fairfax, Virginia
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Ciudad Autonoma de Bueno
- Australia (8):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Macquarie Park, New South Wales
  - GSK Investigational Site, Gold Coast, Queensland
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Melbourne
- Canada (5):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Finland (4):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Turku
- France (8):
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Villeurbanne
- Germany (4):
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Erbach im Odenwald
  - GSK Investigational Site, München
  - GSK Investigational Site, Münster
- Italy (8):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, CefalU PA
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Perugia
- Netherlands (3):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Zwolle
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Stavanger
- South Korea (2):
  - GSK Investigational Site, Junggu
  - GSK Investigational Site, Seoul
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Getxo - Vizcaya
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Terrassa - Barcelona
  - GSK Investigational Site, Valencia
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Tau-Yuan
- Turkey (Türkiye) (2):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, CapaIstanbul
- United Kingdom (4):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/